CLINICAL TRIAL: NCT03273699
Title: Evaluating the Use of Mindfulness Meditation Utilizing a Consumer-Grade EEG Biofeedback Device for Patients Awaiting Treatment for Obsessive Compulsive Disorder
Brief Title: Mindfulness Meditation Utilizing an EEG Biofeedback Device for the Treatment for Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 196-2016
Record Dates: First submitted 2017-08-31; First posted 2017-09-06 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: A repeated measures multivariate analysis of variance (MANOVA) will be conducted with the two groups (guided mindfulness meditation or control wait list group) as the between-group variable and OCD symptom scores as the dependent variables. A mediation analysis will examine whether obsessive beliefs, engagement in thought control strategies, psychological flexibility, and mind wandering mediates treatment related changes in OCD symptom scores (YBOCS, OCI). Daily practice data from the EEG headsets will be automatically uploaded to an encrypted server. These data will be made anonymous from the start of the study; subjects will be identified using their subject I.D. EEG data will be preprocessed and analyzed using EEG Lab (Delorme & Makeig, 2004).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): The study will be a randomized trial where subjects (N=100) will be randomly assigned to receive either 1) an eight week meditation program involving use of an EEG-based biofeedback device, or 2) wait list as per usual. The experimental design is a 2 (treatment condition: Group 1: Mindfulness, Group 2: Control) by 3 (assessment phase: baseline (week 0), mid-treatment (week 4), post-treatment (week 8)) repeated measures factorial design. Group randomization will be completed by the principal investigator, using the "GraphPad Quick Calcs" online calculator which offers simple random allocation into equal-sized groups
  Interventions: Device: Mindfulness
- Control (No Intervention): The study will be a randomized trial where subjects (N=100) will be randomly assigned to receive either 1) an eight week meditation program involving use of an EEG-based biofeedback device, or 2) wait list as per usual. The experimental design is a 2 (treatment condition: Group 1: Mindfulness, Group 2: Control) by 3 (assessment phase: baseline (week 0), mid-treatment (week 4), post-treatment (week 8)) repeated measures factorial design. Group randomization will be completed by the principal investigator, using the "GraphPad Quick Calcs" online calculator which offers simple random allocation into equal-sized groups

INTERVENTIONS:
Device: Mindfulness — Clients will use a consumer grade EEG device that provides guided mindfulness home practices
  Arms: Mindfulness

SUMMARY:
The Frederick W. Thompson Anxiety Disorders Centre has experienced significant demand for services related to the treatment of Obsessive Compulsive Disorder (OCD), resulting in a significant wait time for service. Although Cognitive Behavior Therapy (CBT) is the most efficacious treatment intervention for OCD, there is a growing literature indicating the mindfulness based approaches can be beneficial in terms of managing acute mood and anxiety symptoms as well as reducing relapse risk following treatment.The goal of this study is to examine the potential benefits of using a consumer grade EEG-based biofeedback device that allows clients to engage in home based mindfulness meditation practices while they are waiting to receive clinical services. Specifically, this study will investigate the effects of meditation home practice on symptom alleviation, as related to specific OCD related cognitive processes.

DETAILED DESCRIPTION:
The goal of this study is to examine the potential benefits of using a consumer grade EEG-based biofeedback device that allows clients to engage in home based mindfulness meditation practices while they are waiting to receive clinical services. Specifically, this study will investigate the effects of meditation home practice on symptom alleviation, as related to specific OCD related cognitive processes.The study will be a randomized trial where subjects (N=100) will be randomly assigned to receive either 1) an eight week meditation program involving use of an EEG-based biofeedback device, or 2) wait list as per usual. The experimental design is a 2 (treatment condition: Group 1: Mindfulness, Group 2: Control) by 3 (assessment phase: baseline (week 0), mid-treatment (week 4), post-treatment (week 8)) repeated measures factorial design. Group randomization will be completed by the principal investigator, using the "GraphPad Quick Calcs" online calculator which offers simple random allocation into equal-sized groups.Outcome measures will involve ratings of OCD symptom severity, OCD beliefs, mindfulness, and use of thought control strategies. At baseline, mid treatment (session 4), and post intervention, participants will complete the Yale-Brown Obsessive Compulsive Scale, Obsessive Compulsive Inventory, Obsessive Beliefs Questionnaire, Five Factor Mindfulness Questionnaire, Thought Control Questionnaire, Acceptance and Action Questionnaire, Mind Wandering Scale and the Metacognitions Questionnaire. Once per week, participants will complete the YBOCS, TCQ, and MW. This weekly data will be collected online using the "Survey Monkey" web portal. Daily practice data from the EEG headsets will be automatically uploaded to an encrypted server.

ELIGIBILITY:
Inclusion Criteria:

* All inclusion and exclusion criteria are consistent with the established guidelines for our service - there are no additional study specific criteria. Potential subjects are referred to the service with a query of OCD. Due to the nature of the assessment procedures, which include English-language self-report questionnaires and scales, the ability to communicate in written and spoken English is an inclusion criterion. disorder

Exclusion Criteria:

* Exclusion criteria include a) those with active substance abuse/dependence, b) suspected organic pathology, c) recent suicide attempt/active suicidality, d) active bipolar, psychotic disorder or post-traumatic stress

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (YBOCS) | Completed once per week, for eight weeks
  A self-report inventory of obsessive compulsive symptoms

SECONDARY OUTCOMES:
Obsessive Compulsive Inventory | Completed at three timepoints - week 1, week 4, week 8
  Self-report measure of obsessive compulsive symptoms
Obsessive Beliefs Questionnaire | Completed at three timepoints - week 1, week 4, week 8
  Self-report measure of OCD beliefs
Five Factor Mindfulness Questionnaire | Completed at three timepoints - week 1, week 4, week 8
  Self-report measure of mindfulness
Thought Control Questionnaire | Completed at three timepoints - week 1, week 4, week 8
  Self-report measure of use of thought control strategies
Acceptance and Action Questionnaire | Completed at three timepoints - week 1, week 4, week 8
  Self-report measure of experiential avoidance
Mind Wandering Scale | Completed at three timepoints - week 1, week 4, week 8
  Self-report measure of mind wandering
Metacognitions Questionnaire | Completed at three timepoints - week 1, week 4, week 8
  Self-report measure of metacognitive strategies

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Richter, M.D., Study Director — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhayee S, Tomaszewski P, Lee DH, Moffat G, Pino L, Moreno S, Farb NA. Attentional and affective consequences of technology supported mindfulness training: a randomised, active control, efficacy trial. BMC Psychol. 2016 Nov 29;4(1):60. doi: 10.1186/s40359-016-0168-6. PMID 27894358

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT03273699/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT03273699/ICF_001.pdf